CLINICAL TRIAL: NCT02570763
Title: Combining Non-Invasive Brain Stimulation With Cognitive Behavioral Intervention in Substance Use Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The co-investigator and recipient of funding for the project left the department and we were unable to complete the study without her as a co-investigator.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1508M77345
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Active tDCS; Sham tDCS
Keywords: neurostimulation; comorbidity; tDCS; CBT; anxiety; alcohol
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Stimulation (Experimental): Active tDCS administration during the first 20 minutes of each of the six therapy sessions.
  Interventions: Device: Active tDCS stimulation
- Sham Stimulation (Sham Comparator): Sham tDCS administration during the first 20 minutes of each of six therapy sessions.
  Interventions: Device: Sham tDCS stimulation

INTERVENTIONS:
Device: Active tDCS stimulation
  Arms: Active Stimulation
Device: Sham tDCS stimulation
  Arms: Sham Stimulation

SUMMARY:
The current study aims to examine the safety and feasibility of utilizing tDCS to enhance affect-laden episodic memory consolidation among adults with co-occurring alcohol use and anxiety disorders who have recently undergone detoxification as a step toward the translational clinical application of this approach.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV diagnosis of panic disorder (with or without agoraphobia), generalized anxiety disorder, or social anxiety disorder within the past 30 days
* DSM IV diagnosis of alcohol dependence within the last 30 days
* inpatient treatment at Lodging Plus primarily for alcohol (vs. other drug) dependence
* alcohol use in the 30 days preceding the study
* willingness to provide informed consent
* minimum of a sixth grade English reading level (deemed necessary to complete study materials); as determined by their being able to read and understand the consent form.
* Living within reasonable driving distance (1 hour or less) of the Twin Cities to allow for in-person follow-up interviews

Exclusion Criteria:

* lifetime history of psychosis or mania by history.
* cognitive (e.g., dementia) or physical impairment (e.g., blindness) that interferes with study participation report or as judged by PI/study physician.
* Current suicide risk as deemed by the PI and study physician to be serious and ongoing
* any medical condition or treatment with neurological sequelae (e.g., stroke, tumor, loss of consciousness of more than 30 minutes, HIV, seizures)
* history of ECT
* document loss of consciousness (LOC) for longer than 30 minutes or LOC with neurological sequelae
* pregnancy
* Although seizures are not a known risk of tDCS intervention (Fregni et al., 2006; Nitsche et al., 2008), anyone with a history or a risk for seizures will be excluded from the study
* anyone with metal objects implanted in their head or neck
* anyone taking stimulant medications for any reason as we wish to avoid two sorces of neurostimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Therapy Content Memory Assessment | 24 hours
  Participant's will complete daily assessments of their memory for therapy content from the previous session.